CLINICAL TRIAL: NCT02284009
Title: Study 110933: Albiglutide Versus Placebo in Insulin-treated Subjects With New-onset Type 1 Diabetes Mellitus
Brief Title: Albiglutide Versus Placebo in Insulin-treated Subjects With New-onset Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 110933
Record Dates: First submitted 2014-09-18; First posted 2014-11-05 (Estimated); Results first posted 2019-03-25 (Actual); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: New-onset type 1 diabetes mellitus; Albiglutide
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Albiglutide (Experimental): Approximately 51 subjects will be assigned to albiglutide 30 mg weekly (with treatment-masked increase to 50 mg weekly at Week 6) + background insulin. The starting dose of albiglutide will be 30 mg once weekly and will be increased at Week 6 to 50 mg, once weekly, if the 30-mg weekly dose is tolerated.
  Interventions: Biological: Albiglutide weekly injection; Biological: Insulin
- Placebo (Experimental): Approximately 17 subjects will be assigned to albiglutide matching placebo + background insulin
  Interventions: Biological: Placebo weekly injection; Biological: Insulin

INTERVENTIONS:
Biological: Albiglutide weekly injection — Albiglutide will be provided as a fixed-dose, fully disposable pen injector system having a prefilled dual chamber glass cartridge. To be self-administered as a subcutaneous (SC) injection in the abdomen, thigh or upper arm region. The pen will deliver either 30 mg of albiglutide, 50 mg of albiglutide in a 0.5-mL injection volume. It may be administered at any time of day without regard to meals. It will be administered once a week on the same day each week
  Arms: Albiglutide
Biological: Placebo weekly injection — Placebo provided as a fixed-dose, fully disposable pen injector system having a prefilled dual chamber glass cartridge. To be self-administered as a SC injection in the abdomen, thigh or upper arm region. It may be administered at any time of day, once a week on the same day each week, without regard to meals.
  Arms: Placebo
Biological: Insulin — Commercially available basal/bolus insulin regimen, self administered by the subject, in accordance to the prescription of the physician and as per the package insert

SUMMARY:
This is a Phase II, randomized, double-blind, parallel group, placebo controlled, multicentre study of 52 weeks treatment duration. The primary objective is to evaluate the efficacy(on endogenous insulin secretion), safety and tolerability of weekly albiglutide (a glucagon-like peptide-1 receptor (GLP-1R) agonist) versus placebo when added to insulin therapy in subjects with new-onset type 1 diabetes mellitus (NOT1DM) and residual insulin production.. Approximately 68 eligible subjects will be randomised in a 3:1 ratio such that 51 subjects receive albiglutide 30 milligram (mg) once weekly (with increase to 50 mg once weekly at Week 6 if the 30-mg weekly dose is tolerated) added-on to insulin therapy and 17 subjects receive placebo once weekly added-on to insulin therapy. The total duration of a subject's participation will be approximately 72 weeks (up to 8 weeks of Screening, 52 weeks of treatment and 12 weeks of Post-treatment Follow-up)

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18 to 30 years, inclusive, with a diagnosis of T1DM with an interval of 28-56 days between the initial diagnosis and the first dose of study drug. Documentation of the diagnosis of T1DM (and not just insulin deficiency), including the date of diagnosis, must be obtained from the diagnosing physician.
* Currently requires insulin for T1DM treatment, or has required insulin therapy for T1DM (for >=7 days) between the date of diagnosis and the first dose of study drug. Note: subjects currently taking twice daily commercially available pre-mixed insulin will not be eligible.
* Positive for at least one of the following autoantibodies typically associated with T1DM: antibody to glutamic acid decarboxylase (anti-GAD) antibody to protein tyrosine phosphatase-like protein (anti-IA-2) or an insulin autoantibody (IAA). Please note: A subject who is positive for IAA and negative for the other autoantibodies will not be eligible if the subject has been using insulin for a total of >=7days.
* Evidence of residual functioning pancreatic beta-cells as measured by a peak stimulated C-peptide level > 0.20 nanomoles/litres (nmol/L) during the Screening MMTT when plasma glucose level is >3.9 mmol/L (70 mg/dL) and <=11.1 mmol/L (200 mg/dL). Note: the Screening MMTT should not be performed within one week of resolution of a DKA event.
* Body mass index <=32.0 kilogram/square meters (kg/m^2).
* Female subjects of childbearing potential (i.e., not surgically sterile and/or not postmenopausal) must be practicing adequate contraception (i.e., meeting one of the criteria defined below) from at least 14 days prior to the first dose of randomised study medication until the 12-week post-treatment Follow-up visit : Abstinence from penile-vaginal intercourse, when this is the female's preferred and usual lifestyle; Oral Contraceptive, either combined or progestogen alone ; Injectable progestogen; Implants of etonogestrel or levonorgestrel; Estrogenic vaginal ring; Percutaneous contraceptive patches; Intrauterine device or intrauterine system that has a failure rate of less than 1% per year when used consistently and correctly as stated in the product label; Male partner sterilization prior to the female subject's entry into the study, and this male is the sole partner for that subject. The information on the male sterility can come from the site personnel's review of subject's medical records; medical examination of the subject and/or semen analysis; or interview with the subject on his medical history.; Male condom combined with a female diaphragm, either with or without a vaginal spermicide
* Able and willing to provide written informed consent and to comply with all study procedures.

Exclusion Criteria:

* Severe gastroparesis i.e., requiring therapy within 6 months prior to Screening
* History of acute or chronic pancreatitis, or considered clinically at significant risk of developing pancreatitis, during the course of the study (e.g. due to symptomatic gallstones, excess alcohol use).
* History of significant gastrointestinal surgery that in the opinion of the investigator is likely to significantly affect upper gastrointestinal or pancreatic function (e.g. gastric bypass and banding, antrectomy, Roux-en-Y bypass, gastric vagotomy, small bowel resection, or surgeries thought to significantly affect upper gastrointestinal function)
* Personal history or family history of thyroid medullary carcinoma or multiple endocrine neoplasia type 2 (MEN2)
* History of cancer that has not been in full remission for at least 3 years before Screening. (A history of squamous cell or basal cell carcinoma of the skin, or treated cervical intraepithelial neoplasia I or cervical intraepithelial neoplasia II is allowed)
* Fasting triglyceride level >750 milligram/decilitre (mg/dL) at Screening. Subjects may be re-tested once during screening, and if the value no longer meets the exclusion criterion, the subject can be randomly assigned to treatment
* Estimated Glomerular Filtration Rate (eGFR) <=30 mL/min/1.73 m^2 (calculated using the Modification of Diet in Renal Disease (MDRD) formula
* Haemoglobinopathy that may affect proper interpretation of HbA1c
* Alanine aminotransferase (ALT) >2.5 × upper limit of normal (ULN) and bilirubin >1.5 × ULN (isolated bilirubin >1.5 × ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%)
* Unstable liver disease (as defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, oesophageal or gastric varices or persistent jaundice), cirrhosis, known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones). [Chronic stable hepatitis B and C are acceptable if subject otherwise meets entry criteria and are not on active antiviral treatment (e.g., presence of hepatitis B surface antigen or positive hepatitis C test result within 3 months of screening)]
* Any clinically significant co-morbidity or abnormality (including psychiatric disorder, any other autoimmune endocrinopathy e.g., primary autoimmune hypothyroidism, hyperadrenalism, coeliac disease etc) that in the opinion of the Investigator, may pose additional risk in administering study medication or trial participation
* Female subject is pregnant (confirmed by laboratory testing) or lactating
* Known allergy to any GLP-1 analogue, insulin, or excipients of albiglutide
* Treatment with any oral anti-diabetic medication within the prior 30 days or 5 half lives of that medication, whichever is longer.
* Use of immunosuppressants, intravenous immunoglobulin, oral or systemically injected glucocorticoids within the 3 months before randomisation or high likelihood of a requirement for prolonged treatment (>1 week) in the year following randomisation. However, short courses of oral steroids (single dose or multiple doses for up to 7 days) may be permitted provided these cases are discussed with the medical monitor. Inhaled, intra-articular, and small quantities of non-potent topical corticosteroids are allowed
* Receipt of any investigational drug within the 30 days or 5 half-lives, whichever is longer, before Screening, a history of receipt of an investigational anti-diabetic drug within the 3 months before randomisation, or receipt of albiglutide in previous studies.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2014-10-10 (Actual); Primary Completion 2017-10-18 (Actual); Study Completion 2017-10-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (32):
- France (3):
  - GSK Investigational Site, Bois-Guillaume
  - GSK Investigational Site, Caen
  - GSK Investigational Site, Lille
- Germany (4):
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Düsseldorf, North Rhine-Westphalia
  - GSK Investigational Site, Dresden, Saxony
- Italy (3):
  - GSK Investigational Site, Latina, Lazio
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Roma
- Spain (11):
  - GSK Investigational Site, Alzira/Valencia
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Granada
  - GSK Investigational Site, L'Hospitalet de Llobregat
  - GSK Investigational Site, Lleida
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Pama de Mallorca
  - GSK Investigational Site, San Juan (Alicante)
  - GSK Investigational Site, Seville
- United Kingdom (11):
  - GSK Investigational Site, Birmingham
  - GSK Investigational Site, Bristol
  - GSK Investigational Site, Cardiff
  - GSK Investigational Site, Darlington
  - GSK Investigational Site, Dundee
  - GSK Investigational Site, Durham
  - GSK Investigational Site, Glasgow
  - GSK Investigational Site, Liverpool
  - GSK Investigational Site, London
  - GSK Investigational Site, Newcastle upon Tyne
  - GSK Investigational Site, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20366

REFERENCES:
- [Background] Pozzilli P, Bosi E, Cirkel D, Harris J, Leech N, Tinahones FJ, Vantyghem MC, Vlasakakis G, Ziegler AG, Janmohamed S. Randomized 52-week Phase 2 Trial of Albiglutide Versus Placebo in Adult Patients With Newly Diagnosed Type 1 Diabetes. J Clin Endocrinol Metab. 2020 Jun 1;105(6):dgaa149. doi: 10.1210/clinem/dgaa149. PMID 32219329

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multicenter study conducted at 29 sites in Europe (Spain 10, United Kingdom (UK) 9, Germany 4, France 3 and Italy 3). A total of 67 participants with New-onset type 1 diabetes mellitus (NOT1DM) were randomized.
Pre-assignment Details: Study was terminated early as part of the decision to withdraw albiglutide for commercial reasons. Study stopped after 67 participants were randomized instead of 68 as per protocol. Impact of early termination was minimal and did not affect the interpretation of results.
Groups:
- Placebo: Matching placebo was administered once weekly for 52 weeks by subcutaneous (sc) injection in the abdomen, thigh or upper arm region in addition to insulin.
- Albiglutide: Albiglutide 30 milligram (mg) was administered once weekly for 52 weeks by sc injection in the abdomen, thigh or upper arm region along with insulin (Dose increased to 50 mg once weekly at Week 6 if the 30 mg weekly dose was tolerated).
Period: Overall Study
Arm/Group | Placebo | Albiglutide
Started | 17 | 50
Completed | 11 | 40
Not Completed | 6 | 10
Not completed — Adverse Event | 3 | 0
Not completed — Lost to Follow-up | 1 | 3
Not completed — Physician Decision | 0 | 2
Not completed — Withdrawal by Subject | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Matching placebo was administered once weekly for 52 weeks by sc injection in the abdomen, thigh or upper arm region in addition to insulin.
- Albiglutide: Albiglutide 30 mg was administered once weekly for 52 weeks by sc injection in the abdomen, thigh or upper arm region along with insulin (Dose increased to 50 mg once weekly at Week 6 if the 30 mg weekly dose was tolerated).
- Total: Total of all reporting groups
Arm/Group | Placebo | Albiglutide | Total
Number analyzed (Participants) | 17 | 50 | 67
Age, Continuous [Mean (Standard Deviation); unit: Years] | 22.8 (3.83) | 22.7 (3.72) | 22.7 (3.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 21 | 28
  Male | 10 | 29 | 39
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 0 | 1 | 1
  White | 17 | 49 | 66

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Time Normalized Stimulated (From Mixed Meal Tolerance Test [MMTT]) 2-hour Plasma C-peptide Area Under the Curve (AUC) at Week 52
Description: Participants (parts) had a balanced diet consistent with dietitian's advice and made no major changes in exercise regimens. Evening before the MMTT, participants had a full meal then fasted from 9 post meridiem (pm) until MMTT was completed. Water, black coffee or tea without sugar or artificial sweeteners was allowed. Plasma glucose was measured prior to the finger-stick test and MMTT was performed only if in range > 3.9 millimoles per liter (mmol/L) [70 mg/deciliter (dL)] and <= 11.1 mmol/L (200 mg/dL). Baseline was defined as the last non-missing value with assessment date on or before the 1st day of study medication. Change from Baseline was calculated by subtracting Baseline value from Week 52 value. Intent-to-treat (ITT) Population comprised of all randomly assigned participants who received at least 1 dose of study medication with at least 1 post-Baseline assessment of the primary endpoint.
Time Frame: Baseline and Week 52
Population: ITT Population. Only those participants with available data at the specified time points were analyzed. Time normalized plasma C-peptide AUC was calculated using trapezoidal rule then dividing by 120 (if the result at t=120 is non-missing otherwise the time difference between first and last times with non-missing results is used)
Measure: Mean (Standard Deviation); unit: Nanomoles per liter
Groups:
- DEFEND-1 Placebo: Historical placebo data from the DEFEND-1 (NCT00678886) study was used as prior knowledge.
Arm/Group | Placebo | Albiglutide | DEFEND-1 Placebo
Number analyzed (Participants) | 11 | 40 | 53
Nanomoles per liter | -0.16 (0.366) | -0.13 (0.244) | -0.27 (0.314)
Statistical Analysis 1: Comparison: Placebo vs Albiglutide; Test type: Superiority; Mean Difference (Final Values) = 0.12, 95% CI 2-sided [0.00 to 0.24] — Analysis was performed using a Bayesian model incorporating historical placebo data using a robust mixture prior. Values above are 95% credible intervals. Probability of treatment difference (Albiglutide - Placebo) >= 0.2 nmol/L = 0.097

2. Secondary Outcome: Mean Change From Baseline in Time Normalized Stimulated (From MMTT) 2 Hour Plasma C-peptide AUC at Week 16, 28 and Week 64
Description: Participants had a balanced diet consistent with dietitian's advice and made no major changes in exercise regimens. On the evening before the MMTT, participants had a full meal and then fasted from 9 pm until the MMTT was completed. Water, black coffee or tea without sugar or artificial sweeteners was allowed. Plasma glucose was measured prior to the test using a finger-stick test and MMTT was performed only if it was in range > 3.9 mmol/L (70 mg/dL) and <= 11.1 mmol/L (200 mg/dL). Baseline was defined as the last non-missing value with an assessment date on or before the first day of study medication. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline and Weeks 16, 28 and 64
Population: ITT Population. Only parts with data available at specified data points were analyzed (represented by n= X in the category titles).Time normalized plasma C-peptide AUC was calculated using trapezoidal rule then dividing by 120 (if result at t=120 is non-missing otherwise time difference between first and last times with non-missing results is used)
Measure: Mean (Standard Deviation); unit: Nanomoles per liter
Arm/Group | Placebo | Albiglutide
Number analyzed (Participants) | 15 | 46
Nanomoles per liter
  Week 16, n=15,44: number analyzed (Participants) | 15 | 44
  Week 16, n=15,44 | 0.00 (0.216) | 0.07 (0.234)
  Week 28, n=13,41: number analyzed (Participants) | 13 | 41
  Week 28, n=13,41 | -0.14 (0.177) | 0.01 (0.225)
  Week 64, n=11,36: number analyzed (Participants) | 11 | 36
  Week 64, n=11,36 | -0.22 (0.277) | -0.22 (0.246)

3. Secondary Outcome: Maximum Stimulated Plasma C-peptide (MMTT) at Baseline, Week 16, 28, 52 and 64
Description: Maximum stimulated plasma C-peptide was the highest value at any time point during the 2 hour MMTT after the participant has ingested the mixed meal at Baseline, Week 16, Week 28, Week 52 and Week 64. Blood samples were taken to assess levels of C-peptide at: 10 minutes before Time 0 (-10 minutes), Immediately before the participant starts drinking the nutritional drink (Time 0) and 15, 30, 60, 90, and 120 minutes after Time 0.
Time Frame: Baseline and Weeks 16, 28, 52 and 64
Population: ITT Population. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Measure: Mean (Standard Deviation); unit: Nanomoles per liter
Arm/Group | Placebo | Albiglutide
Number analyzed (Participants) | 15 | 46
Nanomoles per liter
  Baseline, n=15,46 | 0.86 (0.382) | 0.82 (0.448)
  Week 16, n=15,45: number analyzed (Participants) | 15 | 45
  Week 16, n=15,45 | 0.84 (0.481) | 1.02 (0.558)
  Week 28,n=13,42: number analyzed (Participants) | 13 | 42
  Week 28,n=13,42 | 0.68 (0.442) | 0.91 (0.594)
  Week 52,n=11,41: number analyzed (Participants) | 11 | 41
  Week 52,n=11,41 | 0.63 (0.516) | 0.69 (0.479)
  Week 64, n=11,37: number analyzed (Participants) | 11 | 37
  Week 64, n=11,37 | 0.58 (0.453) | 0.48 (0.363)

4. Secondary Outcome: Mean Change From Baseline in Time Normalized Plasma Glucagon AUC (From MMTT) at Week 16, 28, 52 and 64
Description: Blood samples were taken to assess levels of glucagon at: 10 minutes before Time 0 (-10 minutes), immediately before the participant started drinking the nutritional drink (Time 0) and 15, 30, 60, 90, and 120 minutes after Time 0. Mean change from Baseline in time normalized plasma glucagon AUC (from MMTT) at Week 16, 28, 52 and 64 was reported. Baseline was defined as the last non-missing value with an assessment date on or before the first day of study medication. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline and Weeks 16, 28, 52 and 64
Population: ITT Population. Only parts with data available at specified data points were analyzed (represented by n= X in the category titles). Time normalized plasma glucagon AUC was calculated using trapezoidal rule then dividing by 120 (if result at t=120 is non-missing otherwise time difference between first and last times with non-missing results is used)
Measure: Mean (Standard Deviation); unit: Nanograms per liter
Arm/Group | Placebo | Albiglutide
Number analyzed (Participants) | 15 | 46
Nanograms per liter
  Week 16,n=15,45: number analyzed (Participants) | 15 | 45
  Week 16,n=15,45 | -2.28 (11.221) | -1.10 (4.496)
  Week 28,n=13,43: number analyzed (Participants) | 13 | 43
  Week 28,n=13,43 | -2.97 (11.574) | 3.91 (22.197)
  Week 52,n=11,40: number analyzed (Participants) | 11 | 40
  Week 52,n=11,40 | -0.31 (15.989) | 4.66 (13.628)
  Week 64,n=11,37: number analyzed (Participants) | 11 | 37
  Week 64,n=11,37 | 3.19 (18.279) | 8.82 (17.650)

5. Secondary Outcome: Percentage of Responders at Baseline, Weeks 4, 8, 16, 28, 40, 52 and 64
Description: Responders were defined as participants achieving glycosylated hemoglobin A1c (HbA1c) <= 7.0 percent and mean daily insulin use < 0.5 units per kilograms (kg) per day. Percentages are based on the number of participants with available HbA1c and insulin use data in each treatment group at that visit.
Time Frame: Baseline and Weeks 4, 8, 16, 28, 40, 52 and 64
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Albiglutide
Number analyzed (Participants) | 15 | 46
Percentage of participants
  Baseline, n=15, 46 | 26.7 | 37.0
  Week 4,n=14,42: number analyzed (Participants) | 14 | 42
  Week 4,n=14,42 | 71.4 | 78.6
  Week 8,n=14,46: number analyzed (Participants) | 14 | 46
  Week 8,n=14,46 | 85.7 | 67.4
  Week 16,n=15,45: number analyzed (Participants) | 15 | 45
  Week 16,n=15,45 | 86.7 | 73.3
  Week 28,n=12,42: number analyzed (Participants) | 12 | 42
  Week 28,n=12,42 | 75.0 | 73.8
  Week 40,n=13,40: number analyzed (Participants) | 13 | 40
  Week 40,n=13,40 | 76.9 | 62.5
  Week 52,n=12,41: number analyzed (Participants) | 12 | 41
  Week 52,n=12,41 | 41.7 | 48.8
  Week 64,n=11,38: number analyzed (Participants) | 11 | 38
  Week 64,n=11,38 | 36.4 | 34.2

6. Secondary Outcome: Percentage of Participants Achieving Partial Remission Status (Insulin Dose-adjusted Hemoglobin A1c (IDAA1C)<= 9.0) at Baseline, Week 4, 8, 16, 28, 40, 52 and 64
Description: Participant achieving partial remission status was defined as a participant with IDAA1C <=9.0 . Percentages were based on the number of participants with available IDAA1c data in each treatment group at that visit.
Time Frame: Baseline and Weeks 4, 8, 16, 28, 40, 52 and 64
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Albiglutide
Number analyzed (Participants) | 15 | 46
Percentage of participants
  Baseline, n= 15, 46 | 73.3 | 60.9
  Week 4,n=14,42: number analyzed (Participants) | 14 | 42
  Week 4,n=14,42 | 92.9 | 88.1
  Week 8,n=14,46: number analyzed (Participants) | 14 | 46
  Week 8,n=14,46 | 92.9 | 87.0
  Week 16,n=15,45: number analyzed (Participants) | 15 | 45
  Week 16,n=15,45 | 86.7 | 86.7
  Week 28,n=12,42: number analyzed (Participants) | 12 | 42
  Week 28,n=12,42 | 75.0 | 85.7
  Week 40,n=13,40: number analyzed (Participants) | 13 | 40
  Week 40,n=13,40 | 84.6 | 82.5
  Week 52,n=12,41: number analyzed (Participants) | 12 | 41
  Week 52,n=12,41 | 58.3 | 70.7
  Week 64,n=11,38: number analyzed (Participants) | 11 | 38
  Week 64,n=11,38 | 54.5 | 55.3

7. Secondary Outcome: Change From Baseline in Percent HbA1c at Week 52
Description: Change from Baseline in percent HbA1c was reported. Baseline was defined as the last non-missing value with an assessment date on or before the first day of study medication. Change from Baseline was calculated by subtracting Baseline value from the Week 52 value.
Time Frame: Baseline and Week 52
Population: ITT Population. Only those participants with available data at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | Placebo | Albiglutide
Number analyzed (Participants) | 12 | 43
Percentage of HbA1c | -0.73 (1.033) | -0.59 (1.649)

8. Secondary Outcome: Percent HbA1c Over Time (at Weeks 4, 8, 16, 28, 40, 52 and 64)
Description: Blood samples were collected from participants for analysis of HbA1c at indicated time points and percentage of HbA1c has been calculated for Weeks 4, 8, 16, 28, 40, 52 and 64.
Time Frame: Weeks 4, 8, 16, 28, 40, 52 and 64
Population: ITT Population. Only those participants with data available at the specified time points were analyzed (represented by n=x in the category titles).
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | Placebo | Albiglutide
Number analyzed (Participants) | 15 | 46
Percentage of HbA1c
  Week 4,n=15,43: number analyzed (Participants) | 15 | 43
  Week 4,n=15,43 | 6.29 (0.688) | 6.10 (0.725)
  Week 8,n=15,46 | 5.91 (0.689) | 5.82 (0.725)
  Week 16,n=15,46 | 5.97 (0.801) | 5.78 (0.733)
  Week 28,n=13,43: number analyzed (Participants) | 13 | 43
  Week 28,n=13,43 | 6.03 (0.747) | 6.00 (0.824)
  Week 40,n=13,42: number analyzed (Participants) | 13 | 42
  Week 40,n=13,42 | 6.22 (0.860) | 6.20 (0.894)
  Week 52,n=12,43: number analyzed (Participants) | 12 | 43
  Week 52,n=12,43 | 6.56 (0.950) | 6.58 (1.512)
  Week 64,n=12,40: number analyzed (Participants) | 12 | 40
  Week 64,n=12,40 | 7.12 (1.335) | 6.92 (1.176)

9. Secondary Outcome: Change From Baseline in Mean Daily Insulin Use at Week 4, 8, 16, 28, 40, 52 and 64
Description: The mean daily insulin use value was calculated, in units/kg/day as the sum of average prandial insulin doses and average of basal insulin doses for each participant recorded daily for the 3 days prior to the specified visits, divided by the participant's body weight in kg. Baseline was defined as the last non-missing value with an assessment date on or before the first day of study medication. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline and Weeks 4, 8, 16, 28, 40, 52 and 64
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units/kg/day
Arm/Group | Placebo | Albiglutide
Number analyzed (Participants) | 15 | 46
Units/kg/day
  Week 4,n=14,43: number analyzed (Participants) | 14 | 43
  Week 4,n=14,43 | -0.02 (0.076) | -0.03 (0.093)
  Week 8,n=14,46: number analyzed (Participants) | 14 | 46
  Week 8,n=14,46 | -0.04 (0.105) | -0.02 (0.123)
  Week 16,n=15,45: number analyzed (Participants) | 15 | 45
  Week 16,n=15,45 | -0.05 (0.100) | -0.01 (0.148)
  Week 28,n=12,42: number analyzed (Participants) | 12 | 42
  Week 28,n=12,42 | -0.01 (0.139) | 0.03 (0.145)
  Week 40,n=13,40: number analyzed (Participants) | 13 | 40
  Week 40,n=13,40 | -0.01 (0.151) | 0.03 (0.145)
  Week 52,n=12,41: number analyzed (Participants) | 12 | 41
  Week 52,n=12,41 | 0.04 (0.119) | 0.11 (0.215)
  Week 64,n=11,38: number analyzed (Participants) | 11 | 38
  Week 64,n=11,38 | 0.04 (0.140) | 0.10 (0.187)

10. Secondary Outcome: Number of Events of Participant-reported Significant Hypoglycemia, Occurring > Week 24 and <= Week 52
Description: Significant hypoglycemia was defined as an event with plasma glucose level <= 3.9 mmol/L (<= 70 mg/dL) and/or requiring third party intervention. This corresponds to American Diabetes Association (ADA) category definitions of severe, documented symptomatic, and asymptomatic hypoglycemia. The time period was defined as: > Week 24 to <= Week 52 = Day 169 to Day 364. Number of Events were defined as the total number of significant hypoglycemic events at each level of summarization. Number of events of hypoglycemia with confirmed self plasma glucose monitoring <=3.9 mmol/L and/or requiring third party intervention (i.e., severe, documented symptomatic and asymptomatic hypoglycemic events) occurring >Week 24 and <=Week 52 are presented.
Time Frame: Week 24 to 52
Population: ITT Population. Only those participants with available data at specified time points were analyzed
Measure: Number; unit: Hypoglycemic events
Arm/Group | Placebo | Albiglutide
Number analyzed (Participants) | 13 | 45
Hypoglycemic events
  Any Significant Hypoglycemia | 472 | 1592
  Severe Hypoglycemia | 0 | 0
  Documented Symptomatic Hypoglycemia | 241 | 996
  Asymptomatic Hypoglycemia | 231 | 596

11. Secondary Outcome: Time Spent With Plasma Glucose Level <= 3.9, > 3.9 to <= 10.0, and > 10.0 Measured by 72 Hour Continuous Glucose Monitoring (CGM) at Baseline, Week 28 and 52
Description: Three days before the visit, the participants made an additional visit to the study site to have the CGM fitted/inserted. It was worn for 3 consecutive days and was removed at the scheduled study visit. Whilst wearing the CGM, participants continued to monitor their plasma glucose at least 4 times a day and on one of the days, conducted 7-point glucose profile (Before breakfast, 2 hours after breakfast, Before lunch, 2 hours after lunch, Before dinner, 2 hours after dinner, At bedtime). Time spent with a plasma glucose <=3.9 millimoles per liter (mmol/L), between >3.9 and 10.0 mmol/L, and >10.0 mmol/L, respectively as performed by 72-hour CGM at Baseline, Week 28 and Week 52 was reported.
Time Frame: Baseline and Weeks 28 and 52
Population: ITT Population. Only those participants with available data at the specified time points were analysed (represented by n=X in the category titles).
Measure: Mean (Standard Deviation); unit: hours per day
Arm/Group | Placebo | Albiglutide
Number analyzed (Participants) | 15 | 46
hours per day
  <= 3.9 mmol/L, Baseline,n=14,42: number analyzed (Participants) | 14 | 42
  <= 3.9 mmol/L, Baseline,n=14,42 | 0.80 (1.251) | 0.98 (1.400)
  <= 3.9 mmol/L, Week 28,n=12,36: number analyzed (Participants) | 12 | 36
  <= 3.9 mmol/L, Week 28,n=12,36 | 1.72 (1.248) | 1.38 (1.808)
  <= 3.9 mmol/L, Week 52,n=10,31: number analyzed (Participants) | 10 | 31
  <= 3.9 mmol/L, Week 52,n=10,31 | 1.60 (2.142) | 1.36 (2.405)
  > 3.9 to <= 10.0 mmol/L,Baseline,n=14,42: number analyzed (Participants) | 14 | 42
  > 3.9 to <= 10.0 mmol/L,Baseline,n=14,42 | 20.14 (3.675) | 19.11 (3.732)
  > 3.9 to <= 10.0 mmol/L,Week 28,n=12,36: number analyzed (Participants) | 12 | 36
  > 3.9 to <= 10.0 mmol/L,Week 28,n=12,36 | 18.93 (3.452) | 18.83 (4.009)
  > 3.9 to <= 10.0 mmol/L,Week 52,n=10,31: number analyzed (Participants) | 10 | 31
  > 3.9 to <= 10.0 mmol/L,Week 52,n=10,31 | 17.98 (4.491) | 18.19 (4.772)
  > 10.0 mmol/L, Baseline,n=14,42: number analyzed (Participants) | 14 | 42
  > 10.0 mmol/L, Baseline,n=14,42 | 3.06 (3.560) | 3.90 (3.727)
  > 10.0 mmol/L,Week 28,n=12,36: number analyzed (Participants) | 12 | 36
  > 10.0 mmol/L,Week 28,n=12,36 | 3.35 (3.115) | 3.79 (3.782)
  > 10.0 mmol/L,Week 52,n=10,31: number analyzed (Participants) | 10 | 31
  > 10.0 mmol/L,Week 52,n=10,31 | 4.42 (4.597) | 4.45 (4.781)

12. Secondary Outcome: Number of Hypoglycemic Excursions for Each Participant From 7-Point Glucose Profile at Baseline, Week 28 and 52
Description: A hypoglycemic excursion was defined as an occurrence where the plasma glucose level <=3.9 mmol/L (<=70 mg/dL). At each visit, only evaluable participants, defined as those with >= 4 non-missing glucose values or >= 1 hypoglycemic excursions were included. Number of Hypoglycemic Excursions for each participant from 7-Point Glucose Profile (Before breakfast, 2 hours after breakfast, Before lunch, 2 hours after lunch, Before dinner, 2 hours after dinner, At bedtime) were reported. Baseline was defined as the last non-missing value with an assessment date on or before the first day of study medication.
Time Frame: Baseline and Weeks 28 and 52
Population: ITT Population. Only evaluable participants, as defined in the Measure Description were analysed (represented by n=X in the category titles).
Measure: Mean (Standard Deviation); unit: Hypoglycemic excursions
Arm/Group | Placebo | Albiglutide
Number analyzed (Participants) | 15 | 46
Hypoglycemic excursions
  Bseline,n=15,42: number analyzed (Participants) | 15 | 42
  Bseline,n=15,42 | 0.40 (0.632) | 0.36 (0.656)
  Week 28,n=13,40: number analyzed (Participants) | 13 | 40
  Week 28,n=13,40 | 0.31 (0.630) | 0.28 (0.554)
  Week 52,n=12,40: number analyzed (Participants) | 12 | 40
  Week 52,n=12,40 | 0.25 (0.452) | 0.40 (0.672)

13. Secondary Outcome: Greatest Magnitude of Hypoglycemic Excursions for Each Participant From 7-Point Glucose Profile at Baseline, Week 28 and 52
Description: A hypoglycemic excursion was defined as an occurrence where the plasma glucose level <=3.9 mmol/L (<= 70 mg/dL). At each visit, only evaluable participants, defined as those with >= 4 non-missing glucose values or >= 1 hypoglycemic excursions were included. Greatest hypoglycemic excursion was calculated as 3.9 mmol/L minus the lowest recorded glucose level during the 7-point glucose profile (Before breakfast, 2 hours after breakfast, Before lunch, 2 hours after lunch, Before dinner, 2 hours after dinner, At bedtime). If a participant had data recorded at that visit, but did not have a value <= 3.9 mmol/L, their greatest hypoglycemic excursion were 0 mmol/L for that visit. Baseline was defined as the last non-missing value with an assessment date on or before the first day of study medication.
Time Frame: Baseline and Weeks 28 and 52
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | Albiglutide
Number analyzed (Participants) | 15 | 46
mmol/L
  Baseline,n=15,42: number analyzed (Participants) | 15 | 42
  Baseline,n=15,42 | 0.24 (0.470) | 0.22 (0.597)
  Week 28,n=13,40: number analyzed (Participants) | 13 | 40
  Week 28,n=13,40 | 0.18 (0.359) | 0.08 (0.231)
  Week 52,n=12,40: number analyzed (Participants) | 12 | 40
  Week 52,n=12,40 | 0.22 (0.484) | 0.17 (0.393)

14. Secondary Outcome: Number of Hyperglycemic Excursions for Each Participant From 7-Point Glucose Profile at Baseline, Week 28 and 52
Description: A hyperglycemic excursion is defined as an occurrence where the plasma glucose level > 10.0 mmol/L (> 180 mg/dL). At each visit, only evaluable participants, defined as those with >= 4 non-missing glucose values or >= 1 hyperglycemic excursions were included. Number of Hyperglycemic Excursions for each participant from 7-Point Glucose Profile (Before breakfast, 2 hours after breakfast, Before lunch, 2 hours after lunch, Before dinner, 2 hours after dinner, At bedtime) were reported. Baseline was defined as the last non-missing value with an assessment date on or before the first day of study medication.
Time Frame: Baseline and Weeks 28 and 52
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Hyperglycemic excursions
Arm/Group | Placebo | Albiglutide
Number analyzed (Participants) | 15 | 46
Hyperglycemic excursions
  Baseline,n=15,43: number analyzed (Participants) | 15 | 43
  Baseline,n=15,43 | 0.80 (1.014) | 1.53 (1.502)
  Week 28,n=13,40: number analyzed (Participants) | 13 | 40
  Week 28,n=13,40 | 1.23 (1.301) | 0.73 (0.933)
  Week 52,n=12,40: number analyzed (Participants) | 12 | 40
  Week 52,n=12,40 | 1.17 (1.115) | 1.30 (1.522)

15. Secondary Outcome: Greatest Magnitude of Hyperglycemic Excursions for Each Participant From 7-Point Glucose Profile at Baseline, Week 28 and 52
Description: A hyperglycemic excursion is defined as an occurrence where the plasma glucose level > 10.0 mmol/L (> 180 mg/dL). At each visit, only evaluable participants, defined as those with >= 4 non-missing glucose values or >= 1 hyperglycemic excursions were included. Greatest hyperglycemic excursion was calculated as the largest recorded glucose level during the 7-point glucose profile (before breakfast, 2 hours after breakfast, before lunch, 2 hours after lunch, before dinner, 2 hours after dinner, at bedtime) minus 10.0 mmol/L. If a participant had data recorded at that visit, but does not have a value > 10.0 mmol/L, their greatest hyperglycemic excursion would be 0 mmol/L for that visit. Baseline was defined as the last non-missing value with an assessment date on or before the first day of study medication.
Time Frame: Baseline and weeks 28 and 52
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | Albiglutide
Number analyzed (Participants) | 15 | 46
mmol/L
  Baseline,n=15,43: number analyzed (Participants) | 15 | 43
  Baseline,n=15,43 | 0.94 (1.805) | 2.72 (3.466)
  Week 28,n=13,40: number analyzed (Participants) | 13 | 40
  Week 28,n=13,40 | 2.05 (2.154) | 1.52 (2.493)
  Week 52,n=12,40: number analyzed (Participants) | 12 | 40
  Week 52,n=12,40 | 2.19 (2.823) | 2.42 (3.042)

16. Secondary Outcome: Change From Baseline in Body Weight (Kilograms) at Week 52
Description: Change from Baseline in body weight of participants was reported. Baseline was defined as the last non-missing value with an assessment date on or before the first day of study medication. Change from Baseline was calculated by subtracting the Baseline value from the Week 52 value.
Time Frame: Baseline and Week 52
Population: ITT Population. Only those participants with available data at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Placebo | Albiglutide
Number analyzed (Participants) | 12 | 43
Kilograms | 0.26 (2.738) | 0.77 (3.504)

17. Secondary Outcome: Weight Over Time (at Weeks 2, 4, 6, 8, 16, 28, 40, 52 and 64)
Description: Body weight was measured in kilograms for participants at indicated time points.
Time Frame: Weeks 2, 4, 6, 8, 16, 28, 40, 52 and 64
Population: ITT Population. Only participants with available data at the specified time points were summarized
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Placebo | Albiglutide
Number analyzed (Participants) | 15 | 46
kilograms
  Week 2,n=15, 43: number analyzed (Participants) | 15 | 43
  Week 2,n=15, 43 | 70.16 (14.087) | 66.16 (11.944)
  Week 4,n=15, 44: number analyzed (Participants) | 15 | 44
  Week 4,n=15, 44 | 69.87 (14.409) | 66.39 (11.952)
  Week 6,n=15, 46 | 69.83 (14.013) | 65.65 (12.559)
  Week 8,n=15, 46 | 70.08 (14.121) | 65.32 (12.825)
  Week 16,n=15, 46 | 69.40 (15.191) | 65.41 (12.824)
  Week 28,n=13, 43: number analyzed (Participants) | 13 | 43
  Week 28,n=13, 43 | 66.08 (11.767) | 65.32 (13.252)
  Week 40,n=13, 42: number analyzed (Participants) | 13 | 42
  Week 40,n=13, 42 | 66.08 (11.266) | 66.20 (13.146)
  Week 52,n=12, 43: number analyzed (Participants) | 12 | 43
  Week 52,n=12, 43 | 66.86 (12.401) | 66.80 (12.696)
  Week 64,n=12, 40: number analyzed (Participants) | 12 | 40
  Week 64,n=12, 40 | 68.29 (11.511) | 68.13 (12.649)

18. Secondary Outcome: Population Estimates of Pharmacokinetic (PK) Parameters: Apparent Clearance [CL/F]
Description: PK of Albiglutide was evaluated in participants using CL/F using PK samples collected on Weeks 4, 6, 8, 16. CL/F was evaluated by population PK methods and mean and standard error from the final model has been tabulated. Estimates have been presented from the final model centered to mean body weights of 67 kilograms, and electronic glomerular filtration rate (eGFR) of 123 milliliters per minute.
Time Frame: 48 hours after the most recent dose at Week 4, 6, 8 and 16
Population: PK population which comprised of participants in 'Safety Population' for whom a pharmacokinetic sample was obtained and analyzed. Only participants who received albiglutide were included in PK Population.
Measure: Mean (Standard Error); unit: Milliliters per hour
Arm/Group | Albiglutide
Number analyzed (Participants) | 49
Milliliters per hour | 45.1 (2.56)

19. Secondary Outcome: Population Estimates of PK Parameters: Apparent Volume of Distribution [V/F]
Description: PK of Albiglutide was evaluated in participants using V/F using PK samples collected on Weeks 4, 6, 8, 16. V/F was evaluated by population PK methods and mean and standard error from the final model has been tabulated. Estimates have been presented from the final model centered to mean body weights of 67 kilograms, and eGFR of 123 milliliters per minute.
Time Frame: 48 hours after the most recent dose at Week 4, 6, 8 and 16
Population: PK population
Measure: Mean (Standard Error); unit: Milliliters
Arm/Group | Albiglutide
Number analyzed (Participants) | 49
Milliliters | 4830 (677)

20. Secondary Outcome: Population Estimates of PK Parameters: First-order Absorption Rate Constant [Ka]
Description: PK of Albiglutide was evaluated in participants using Ka using PK samples collected on Weeks 4, 6, 8, 16. Ka was evaluated by population PK methods and mean and standard error from the final model has been tabulated. Estimates have been presented from the final model centered to mean bodyweights of 67 kilograms, and eGFR of 123 milliliters per minute.
Time Frame: 48 hours after the most recent dose at Week 4, 6, 8 and 16
Population: PK population
Measure: Mean (Standard Error); unit: Per hour
Arm/Group | Albiglutide
Number analyzed (Participants) | 49
Per hour | 0.0122 (0.0022)

ADVERSE EVENTS:
Time Frame: On-therapy AEs and SAEs were collected from start of study treatment up to 52-weeks
Description: AEs and SAEs were summarized in Safety Population. Safety Population comprised of all participants who received at least one dose of study treatment.
Arm/Group | Placebo | Albiglutide
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/50
Serious Adverse Events (participants affected / at risk) | 2/17 | 1/50
Other Adverse Events (participants affected / at risk) | 13/17 | 37/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=17) | Albiglutide (N=50)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=17) | Albiglutide (N=50)
Nausea (Gastrointestinal disorders) | 5 | 19
Diarrhoea (Gastrointestinal disorders) | 2 | 13
Vomiting (Gastrointestinal disorders) | 4 | 10
Abdominal distension (Gastrointestinal disorders) | 0 | 7
Abdominal pain (Gastrointestinal disorders) | 0 | 7
Abdominal pain upper (Gastrointestinal disorders) | 3 | 4
Dyspepsia (Gastrointestinal disorders) | 0 | 3
Flatulence (Gastrointestinal disorders) | 1 | 2
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 1
Nasopharyngitis (Infections and infestations) | 5 | 13
Influenza (Infections and infestations) | 0 | 4
Gastroenteritis (Infections and infestations) | 0 | 3
Urinary tract infection (Infections and infestations) | 1 | 2
Folliculitis (Infections and infestations) | 2 | 0
Sinusitis (Infections and infestations) | 1 | 1
Bronchitis (Infections and infestations) | 1 | 0
Candida infection (Infections and infestations) | 1 | 0
Laryngitis (Infections and infestations) | 1 | 0
Paronychia (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Tooth infection (Infections and infestations) | 1 | 0
Varicella (Infections and infestations) | 1 | 0
Headache (Nervous system disorders) | 5 | 4
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Asthenia (General disorders) | 2 | 1
Injection site erythema (General disorders) | 0 | 3
Malaise (General disorders) | 0 | 3
Pyrexia (General disorders) | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 3
Eczema (Skin and subcutaneous tissue disorders) | 1 | 1
Lipodystrophy acquired (Skin and subcutaneous tissue disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2014-09-24): https://cdn.clinicaltrials.gov/large-docs/09/NCT02284009/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-01): https://cdn.clinicaltrials.gov/large-docs/09/NCT02284009/SAP_001.pdf